CLINICAL TRIAL: NCT04458454
Title: "Study of the Effects of Serum and Follicular Fluid Relaxin Levels on Ovarian Function in IVF Cycles as a Part of the Project "Relaxifert" "
Brief Title: "Study of the Effects of Serum and Follicular Fluid Relaxin Levels on Ovarian Function in IVF Cycles"
Acronym: "Relaxifert"
Status: Completed | Type: Observational
Sponsor: D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology (Other)
Responsible Party: Principal Investigator, Olesya Nikolaevna Bespalova, Olesya Nikolaevna Bespalova, MD, PhD, DSci (Medicine), Deputy Director for Research. The Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott, D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Other Study IDs: DOOttResearch
Record Dates: First submitted 2020-05-09; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Infertility; Reproductive Techniques, Assisted; Oocyte Maturation
Keywords: Infertility; Relaxin; Oocytes; Embryo quality; IVF
MeSH Terms: conditions — Infertility; Helping Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Examination of relaxin levels: This is a pilot study of 1 group of patients. The analysis of relaxin levels in serum and follicular fluid obtained on the day of puncture of the follicles in patients undergoing treatment in the IVF protocol is carried out.
  Interventions: Diagnostic Test: Relaxin ELISA Kit

INTERVENTIONS:
Diagnostic Test: Relaxin ELISA Kit — Ovarian stimulation was carried out from day 3 of the menstrual cycle using a fixed protocol, with recombinant (Gonal-F, Pergoveris) or human menopausal gonadotropins (Meriofert), GnRH antagonist (ganirelix 0.25 mg). A recombinant human chorionic gonadotropin Ovitrel 250 μg or a GnRH agonist, Diferelin 0.2 mg, was used as an ovulation trigger.

SUMMARY:
The study evaluated the effect of serum relaxin and follicular fluid levels on the number and quality of oocytes, fertilization, the number and quality of the embryos in IVF protocols.

DETAILED DESCRIPTION:
Relaxin is one of the promising indicators of oocyte quality and prognosis of the effectiveness of invitro fertilization protocols. The hormone plays an important role in the processes of folliculogenesis, growth and maturation of oocytes, development of embryos, implantation processes, pregnancy and childbirth. A pilot study was conducted on a group of patients undergoing infertility treatment using assisted reproductive technologies in the superovulation stimulation protocol using gonadotropin releasing hormone antagonists. Blood and follicular fluid samples were obtained on the day of transvaginal follicular puncture. The results allow us to consider the hormone relaxin as a promising predictor of the result of ovarian stimulation, the effectiveness of fertilization in IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Primary or Secondary infertility
2. Must be signed the voluntary informed consent to participate in the study.

Exclusion Criteria:

1. The presence of IVF contra-indications.
2. Clinical diagnosis of large uterine fibroids.
3. BMI> 35 kg / m2
4. Morphological diagnosis of endometrial hyperplastic processes
5. Clinical diagnosis of infectious.
6. Clinical diagnosis of systemic autoimmune diseases.
7. Insulin dependent diabetes
8. Oncological diseases

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: The study included patients undergoing treatment in the Department of Assisted Reproductive Technologies of The Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott, Saint Petersburg, Russia
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation between the relaxin values in follicular fluid and the number of oocytes obtained | 10-14 days from the start of stimulation in the IVF protocol ( the day of transvaginal follicular puncture)
  The level of relaxin in follicular fluid was estimated using an ELISA Kit for Relaxin 2. The range of detectable concentrations was 3.1-500 pg / ml. Higher relaxin concentrations in follicular fluid are associated with a higher number of oocytes obtained.

SECONDARY OUTCOMES:
Correlation between the relaxin levels in follicular fluid and oocyte fertilization efficiency | 10-14 days from the start of stimulation in the IVF protocol for relaxin. The first day after transvaginal follicular puncture for evaluation oocyte fertilization efficiency.
  The level of relaxin in follicular fluid was estimated using an ELISA Kit for Relaxin 2. The range of detected concentrations was 3.1-500 pg / ml. In course of standard IVF technique the fertilization efficacy was evaluated as a ratio of double pro-nucleus zygote on the 1st day of development to obtained oocyte-cumulus complexes number. In course of ICSI the efficacy was estimated as ratio of double pro-nucleus zygote on the 1st day of development to oocyte number on MII stage on puncture day. Higher concentrations of follicular fluid relaxin are associated with a decrease efficacy of oocyte fertilization
Correlation between the relaxin levels in follicular fluid and age | 10-14 days from the start of stimulation in the IVF protocol
  The method of relaxin determining in follicular fluid and the range of determined concentrations are described previously. With increasing age, a decrease in the concentration of relaxin in the follicular fluid was noted.
Correlation between the relaxin levels in follicular fluid and BMI | 10-14 days from the start of stimulation in the IVF protocol
  The method of relaxin determining in follicular fluid and the range of determined concentrations are described previously. With increasing of BMI, a decrease in the concentration of relaxin in the follicular fluid was noted.

CONTACTS AND LOCATIONS:
Overall Officials: Olesya N Bespalova, MD, DSci, Principal Investigator — D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Locations (1):
- DOOttResearch, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
For this study, do not see the need to publish these data.